CLINICAL TRIAL: NCT01132807
Title: Phase II Trial of Response-Adapted Chemotherapy Based on Positron Emission Tomography for Non-Bulky Stage I and II Hodgkin Lymphoma
Brief Title: Chemotherapy Based on Positron Emission Tomography Scan in Treating Patients With Stage I or Stage II Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50604; CALGB-50604; NCI-2011-02042 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH); CDR0000672913 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Doxorubicin; Procarbazine; Vinblastine; Dacarbazine; Cyclophosphamide; etoposide phosphate; Prednisone; Radiotherapy; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy and F-18 PET/CT) (Experimental): See Detailed Description
  Interventions: Biological: Bleomycin Sulfate; Drug: Doxorubicin Hydrochloride; Drug: Procarbazine Hydrochloride; Drug: Vinblastine Sulfate; Drug: Dacarbazine; Drug: Cyclophosphamide; Drug: Etoposide phosphate; Drug: prednisone; Drug: Radiation Therapy; Radiation: Fludeoxyglucose F-18; Procedure: computed tomography; Procedure: Positron Emission Tomography

INTERVENTIONS:
Biological: Bleomycin Sulfate — Given IV
Drug: Doxorubicin Hydrochloride — Given IV
Drug: Procarbazine Hydrochloride — Given PO
Drug: Vinblastine Sulfate — Given IV
Drug: Dacarbazine — Given IV
Drug: Cyclophosphamide — Given IV
Drug: Etoposide phosphate — Given IV
Drug: prednisone — Given PO
Drug: Radiation Therapy — Undergo radiation therapy
Radiation: Fludeoxyglucose F-18 — Undergo FDG PET/CT
Procedure: computed tomography — Undergo FDG PET/CT
Procedure: Positron Emission Tomography — Undergo FDG PET/CT

SUMMARY:
This phase II trial studies how well chemotherapy based on positron emission tomography (PET) scan works in treating patients with stage I or stage II Hodgkin lymphoma. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Radiation therapy uses high energy x-rays to kill cancer cells. Giving combination chemotherapy together with radiation therapy may kill more cancer cells and allow doctors to save the part of the body where the cancer started. Comparing results of diagnostic procedures, such as PET scan, done before, during, and after chemotherapy may help doctors predict a patient's response to treatment and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the progression-free survival (PFS) from enrollment for patients with non-bulky stage I and II Hodgkin lymphoma.

II. To compare the PFS of patients who are PET positive versus PET negative following 2 cycles of doxorubicin hydrochloride, bleomycin, vinblastine, and dacarbazine (ABVD).

SECONDARY OBJECTIVES:

I. To evaluate the complete response (CR) rate of patients diagnosed with non-bulky stage I and II Hodgkin lymphoma following PET response-adapted chemotherapy with or without radiation therapy.

II. To determine the predictive value of fludeoxyglucose (FDG) uptake using various semi-quantitative approaches, at baseline, after 2 cycles of AVBD and at completion of therapy.

III. To determine the predictive value of volumetric changes on computed tomography (CT) vs 2-dimensional (2-D) analyses after 2 cycles and 4 cycles and compare with PET parameters with and without combination analyses (PET + dedicated CT data).

IV. To compare the predictive value of metabolic parameters/changes that are measured both visually and semi-quantitatively, International Harmonization Project (IHP) criteria, 2-D and volumetric CT changes, molecular parameters, and conventional parameters, including International Prognostic Score (IPS).

V. To assess whether elevated baseline circulating markers of inflammation (including soluble cluster of differentiation CD30 [sCD]30, soluble CD 163 [CD163], interleukin-10 (IL10), chemokine (C-C motif) ligand 17 (CCL17), and chemokine (C-C motif) ligand 22 [CCL22]) correlate with clinical response and PFS and PET scan results.

VI. To assess whether persistent or recurrent elevated serial circulating markers of inflammation (including soluble CD30 [sCD30], soluble CD163 [sCD163], IL10, CCL17, or CCL22) correlate with relapse/progression or PET scan results.

VII. To confirm independently useful tissue biomarkers for risk stratification in patients with non-bulky stage I and II Hodgkin lymphoma treated with this regimen.

VIII. To compare mediastinal bulk on standing posterior-anterior (PA) and lateral chest x-ray (> 0.33 maximum chest diameter) with chest CT (mass > 10 cm).

OUTLINE:

ABVD CHEMOTHERAPY: Patients receive doxorubicin hydrochloride intravenously (IV) over 3-5 minutes, bleomycin sulfate IV over 3-5 minutes, vinblastine IV over 3-5 minutes, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 2 courses. Patients then undergo PET scan. Patients achieving complete response (CR), partial response (PR), or stable disease (SD) with a negative PET scan receive 2 additional courses of ABVD chemotherapy in the absence of disease progression or unacceptable toxicity. Patients achieving CR, PR, or SD with a positive PET scan proceed to escalated BEACOPP chemotherapy.

ESCALATED BEACOPP* CHEMOTHERAPY: Patients receive doxorubicin hydrochloride IV over 3-5 minutes and cyclophosphamide IV over 60 minutes on day 1, etoposide IV over 45-60 minutes on days 1-3, procarbazine orally (PO) on days 1-7, prednisone PO on days 1-14, and bleomycin sulfate IV and vincristine IV on day 8. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Within 4-6 weeks after completion of BEACOPP chemotherapy, patients undergo involved-field radiotherapy (IFRT) 5 days a week for 3½ weeks.

NOTE: * HIV-positive patients receive standard BEACOPP instead of escalated BEACOPP.

Patients undergo fludeoxyglucose F^18 PET/CT scan at baseline, and within 8-10 days after completion of chemotherapy. Patients also undergo additional PET/CT scans within 3-4 weeks after completion of ABVD or within 12 weeks after completion of BEACOPP and IFRT. Patients with a negative PET scan proceed to follow up. Patients with a positive PET scan undergo biopsy**. Patients with a negative biopsy proceed to follow up, and patients with a positive biopsy are treated at the discretion of the investigator.

NOTE: ** Patients for whom biopsy is neither clinically appropriate nor medically feasible proceed to follow-up. Patients for whom biopsy is neither clinically indicated nor medically appropriate undergo a repeat PET/CT scan after 3 months. If PET/CT scan remains positive, patients undergo biopsy as above.

After completion of study therapy, patients are followed up every 3 months for 1 year, every 6 months for 2-3 years, and then annually for a maximum of 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* Hodgkin lymphoma

  * Clinical stage IA, IB, IIA, or IIB disease according to the modified Ann Arbor Staging Classification system
  * Subclassified according to the WHO modification of the Rye Classification
  * "E" extension allowed provided all other criteria have been met NOTE: *Pathology materials must be submitted within 60 days of study registration. Core-needle biopsies are acceptable provided they contain adequate tissue for primary diagnosis and immunophenotyping. Fine-needle aspirates not allowed. If multiple specimens are available, submit the most recent.
* No nodular lymphocyte-predominant Hodgkin lymphoma
* No mediastinal mass > 0.33 maximum intrathoracic diameter by standing postero-anterior chest x-ray or peripheral or retroperitoneal adenopathy > 10 cm in its largest diameter
* Measurable disease by physical examination or imaging studies

  * Any tumor mass measurable in two dimensions and > 1 cm (or 1.5 cm if 0.5 cm slices are used, as in spiral CT scans) allowed
  * Lesions that are considered intrinsically non-measurable include:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Lesions that are situated in a previously irradiated area

PATIENT CHARACTERISTICS:

* Performance status 0-2
* ANC ≥ 1,000/μL
* Platelet count ≥ 100,000/μL
* Serum creatinine ≤ 2 mg/dL
* Bilirubin ≤ 2 mg/dL
* AST ≤ 2 times upper limit of normal
* LVEF normal by ECHO or MUGA
* DLCO ≥ 60% with no symptomatic pulmonary disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients with known HIV allowed provided they have CD4 counts ≥ 350/mcL

  * Patients must not have multi-drug resistant HIV infections (i.e., concurrent AIDS-defining conditions)
  * An HIV test is required for patients with a history of IV drug abuse or any behavior associated with an increased risk of HIVinfection
* No "currently active" second malignancy other than nonmelanoma skin cancers

  * Patients are not considered to have a "currently active" malignancy provided they have completed therapy and are considered by their physician to be at < 30% risk of relapse

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy for Hodgkin lymphoma

  * 1 course of ABVD (doxorubicin, bleomycin, vinblastine, and dacarbazine) allowed and will be considered the first course

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2010-05; Primary Completion 2016-02 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Straus, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (95):
- United States (95):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Yale Cancer Center, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - McFarland Clinic, PC, Ames, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - Norton Suburban Hospital, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Fox Chase Cancer Center CCOP Research Base, Philadelphia, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Straus DJ, Jung SH, Pitcher B, Kostakoglu L, Grecula JC, Hsi ED, Schoder H, Popplewell LL, Chang JE, Moskowitz CH, Wagner-Johnston N, Leonard JP, Friedberg JW, Kahl BS, Cheson BD, Bartlett NL. CALGB 50604: risk-adapted treatment of nonbulky early-stage Hodgkin lymphoma based on interim PET. Blood. 2018 Sep 6;132(10):1013-1021. doi: 10.1182/blood-2018-01-827246. Epub 2018 Jul 26. PMID 30049811

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Therapy consisted of 2-28 day cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle. PET/CT central review occurred after cycle 2. PET-negative patients received 2 additional cycles of ABVD. PET-positive patients received 2-21 day cycles of 3060-cGy involved-field RT (IFRT) and escalated BEACOPP.
Groups:
- Only Initial ABVD Treatment: Therapy consisted of 2 initial cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle. A cycle is 28 days.>
  * Doxorubicin 25 mg/m2 IV on Days 1 and 15>
  * Bleomycin 10 units/m2 IV on Days 1 and 15>
  * Vinblastine 6 mg/m2 IV on Days 1 and 15>
  * Dacarbazine 375 mg/m2 IV infusion on Days 1 and 15
- Treatment (ABVD:Additional 2 Cycles): Therapy consisted of an initial 2-28 day cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle. A cycle is 28 days.>
  * Doxorubicin 25 mg/m2 IV on Days 1 and 15>
  * Bleomycin 10 units/m2 IV on Days 1 and 15>
  * Vinblastine 6 mg/m2 IV on Days 1 and 15>
  * Dacarbazine 375 mg/m2 IV infusion on Days 1 and 15>
  Patients underwent a PET/CT central review (cycle 2, days 23-25) and received an additional 2-28 day cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle.
- Escalated BEACOPP and Involved Field Radiation Therapy: Therapy consisted of 2-28 day cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle. >
  * Doxorubicin 25 mg/m2 IV on Days 1 and 15>
  * Bleomycin 10 units/m2 IV on Days 1 and 15>
  * Vinblastine 6 mg/m2 IV on Days 1 and 15>
  * Dacarbazine 375 mg/m2 IV infusion on Days 1 and 15> >> > >> Patients underwent a PET/CT central review (cycle 2, days 23-25) and received an additional 2-21 day cycles of 3060-cGy involved-field RT (IFRT) and escalated BEACOPP:> >> > >> Bleomycin 10 units/m2 IV on Day 8> >> Etoposide 200 mg/m2 IV over 60 minutes on Days 1, 2 and 3 > >> Doxorubicin 35 mg/m2 IV on Day 1 > >> Cyclophosphamide 1250 mg/m2 IV over 60 minutes on Day 1 > >> Vincristine 1.4 mg/m2 (maximum 2 mg) IV on Day 8 > >> Procarbazine 100 mg/m2 (rounded to nearest 50 mg) orally on Days 1-7>
  Prednisone 40 mg/m2 (rounded to nearest 5 mg) orally on Days 1-14
Period: Initial ABVD Treatment (2 Cycles)
Arm/Group | Only Initial ABVD Treatment | Treatment (ABVD:Additional 2 Cycles) | Escalated BEACOPP and Involved Field Radiation Therapy
Started | 15 | 135 | 14
Completed | 0 | 135 | 14
Not Completed | 15 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Not completed — Ineligible | 6 | 0 | 0
Period: Post-Cycle 2 PET Assessment
Arm/Group | Only Initial ABVD Treatment | Treatment (ABVD:Additional 2 Cycles) | Escalated BEACOPP and Involved Field Radiation Therapy
Started | 0 | 135 | 14
Completed | 0 | 135 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that began protocol treatment and were eligible for inclusion in any endpoint analysis are included in baseline characteristics.
Groups:
- Treatment (ABVD x2 Cycles): Therapy consisted of 2 cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle. A cycle is 28 days.>>
  * Doxorubicin 25 mg/m2 IV on Days 1 and 15>>
  * Bleomycin 10 units/m2 IV on Days 1 and 15>>
  * Vinblastine 6 mg/m2 IV on Days 1 and 15>>
  * Dacarbazine 375 mg/m2 IV infusion on Days 1 and 15>> >> PET/CT central review (cycle 2, days 23-25). Patients with a negative PET/CT (Deauville 1, 2, or 3) received 2 additional cycles of ABVD. >> >> Patients with positive PET received 2-21 day cycles of 3060-cGy involved-field RT (IFRT) and escalated BEACOPP:>>
  Bleomycin 10 units/m2 IV on Day 8>> Etoposide 200 mg/m2 IV over 60 minutes on Days 1, 2 and 3 >> Doxorubicin 35 mg/m2 IV on Day 1 >> Cyclophosphamide 1250 mg/m2 IV over 60 minutes on Day 1 >> Vincristine 1.4 mg/m2 (maximum 2 mg) IV on Day 8 >> Procarbazine 100 mg/m2 (rounded to nearest 50 mg) orally on Days 1-7>> Prednisone 40 mg/m2 (rounded to nearest 5 mg) orally on Days 1-14
Arm/Group | Treatment (ABVD x2 Cycles)
Number analyzed (Participants) | 164
Age, Continuous [Median (Full Range); unit: years] | 31 [18 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 88
Region of Enrollment [Number; unit: participants]
  United States | 164

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) at 36-Months for Patients Who Received 4 Cycles of ABVD
Description: The primary objective of this trial is to estimate the 3 year PFS in patients who received 4 cycles of ABVD. PFS for each patient is measured as the time from registration on trial to the first incident of death or progression. The PFS at 36 months is calculated as the number of patients who have a progression-free survival time greater than 36 months divided by the total number of patients that started treatment. For this endpoint, all patients that received 4 cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) are included.
Time Frame: 36 Months
Population: All patients that received 4 cycles of ABVD were included in this analysis
Measure: Number (95% Confidence Interval); unit: proportion of patients
Groups:
- Treatment (ABVD: 4 Cycles): Therapy consisted of 2-28 day cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle. A cycle is 28 days.
  * Doxorubicin 25 mg/m2 IV on Days 1 and 15
  * Bleomycin 10 units/m2 IV on Days 1 and 15
  * Vinblastine 6 mg/m2 IV on Days 1 and 15
  * Dacarbazine 375 mg/m2 IV infusion on Days 1 and 15
  PET/CT central review (cycle 2, days 23-25). Patients with a negative PET/CT (Deauville 1, 2, or 3) received 2 additional cycles of ABVD.
Arm/Group | Treatment (ABVD: 4 Cycles)
Number analyzed (Participants) | 135
proportion of patients | .91 [.84 to .95]

2. Primary Outcome: 36 Month Progression Free Survival Rate of Patients Receiving 4 Cycles of ABVD Versus Patients Receiving 2 Cycles of ABVD and 2 Cycles of BEACOPP and Radiation.
Description: All patients received an initial 2-28 day cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15. After the first 2 cycles of ABVD, PET/CT was performed and submitted for central review (cycle 2, days 23-25) and determined whether patients would receive 2 cycles of escalated BEACOPP and involved-field RT (IFRT) or an additional 2 cycles of ABVD. PFS for each patient is measured as the time from registration on trial to the first incident of death or progression. The PFS rate at 36 months is calculated as the number of patients who have a progression-free survival time greater than 36 months divided by the total number of patients that started treatment. For this endpoint, we compare the PFS rate between patients who received 4 cycles of ABVD and patients who received 2 cycles of ABVD and 2 cycles of IFRT.
Time Frame: at 36 months
Population: All patients that completed an initial 2 cycles of ABVD were included in this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Treatment (ABVD:4 Cycles): Therapy consisted of 2-28 day cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle. A cycle is 28 days.
  * Doxorubicin 25 mg/m2 IV on Days 1 and 15
  * Bleomycin 10 units/m2 IV on Days 1 and 15
  * Vinblastine 6 mg/m2 IV on Days 1 and 15
  * Dacarbazine 375 mg/m2 IV infusion on Days 1 and 15
  PET/CT central review (cycle 2, days 23-25). Patients with a negative PET/CT (Deauville 1, 2, or 3) received 2 additional cycles of ABVD.
- Escalated BEACOPP and Involved Field Radiation Therapy: Therapy consisted of 2 cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle. A cycle is 28 days.
  * Doxorubicin 25 mg/m2 IV on Days 1 and 15
  * Bleomycin 10 units/m2 IV on Days 1 and 15
  * Vinblastine 6 mg/m2 IV on Days 1 and 15
  * Dacarbazine 375 mg/m2 IV infusion on Days 1 and 15
  PET/CT central review (cycle 2, days 23-25). Patients with positive PET received 2-21 day cycles of 3060-cGy involved-field RT (IFRT) and escalated BEACOPP:
  >
  > Bleomycin 10 units/m2 IV on Day 8
  > Etoposide 200 mg/m2 IV over 60 minutes on Days 1, 2 and 3
  > Doxorubicin 35 mg/m2 IV on Day 1
  > Cyclophosphamide 1250 mg/m2 IV over 60 minutes on Day 1
  > Vincristine 1.4 mg/m2 (maximum 2 mg) IV on Day 8
  > Procarbazine 100 mg/m2 (rounded to nearest 50 mg) orally on Days 1-7
  > Prednisone 40 mg/m2 (rounded to nearest 5 mg) orally on Days 1-14
Arm/Group | Treatment (ABVD:4 Cycles) | Escalated BEACOPP and Involved Field Radiation Therapy
Number analyzed (Participants) | 135 | 14
proportion of participants | .91 [.84 to .95] | .67 [.34 to .86]

3. Secondary Outcome: Complete Response Rate
Description: A Complete Response (CR) was defined as having the following conditions: 1. A complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. 2. In patients with a PET scan that was positive before therapy, a post-treatment residual mass of any size is permitted as long as it is PET-negative. A Complete Response rate was defined as the number of patients who achieved a CR divided by the number of patients that were eligible for analysis in each group. The CR rate was calculated for patients that completed 4 cycles of ABVD and for patients that completed 2 cycles of ABVD and 2 cycles of BEACOPP and IFRT.
Time Frame: Up to 5 years
Population: Two patients began a third cycle of ABVD and were not eligible for response evaluation (one withdrew and one was lost to follow up). Fourteen patients started BEACOPP treatment, and one patient was lost to follow-up and not included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (ABVD: 4 Cycles) | Escalated BEACOPP and Involved Field Radiation Therapy
Number analyzed (Participants) | 133 | 13
proportion of participants | .97 [.94 to 1.00] | .85 [.65 to 1.00]

ADVERSE EVENTS:
Time Frame: Adverse events were collected after every cycle of treatment up to 4 -28 day cycles.
Groups:
- Only Initial Treatment (ABVD x2 Cycles): Prednisone 40 mg/m2 (rounded to nearest 5 mg) orally on Days 1-14
- Treatment (ABVD:4 Cycles): Therapy consisted of 2-28 day cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle. A cycle is 28 days.
  Doxorubicin 25 mg/m2 IV on Days 1 and 15 Bleomycin 10 units/m2 IV on Days 1 and 15 Vinblastine 6 mg/m2 IV on Days 1 and 15 Dacarbazine 375 mg/m2 IV infusion on Days 1 and 15
  PET/CT central review (cycle 2, days 23-25). Patients with a negative PET/CT (Deauville 1, 2, or 3) received 2 additional cycles of ABVD.
- Escalated BEACOPP and Involved Field Radiation Therapy: Therapy consisted of 2 cycles of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) on Days 1 and 15 of each cycle. A cycle is 28 days.
  Doxorubicin 25 mg/m2 IV on Days 1 and 15 Bleomycin 10 units/m2 IV on Days 1 and 15 Vinblastine 6 mg/m2 IV on Days 1 and 15 Dacarbazine 375 mg/m2 IV infusion on Days 1 and 15
  PET/CT central review (cycle 2, days 23-25). Patients with positive PET received 2-21 day cycles of 3060-cGy involved-field RT (IFRT) and escalated BEACOPP:
  Bleomycin 10 units/m2 IV on Day 8 Etoposide 200 mg/m2 IV over 60 minutes on Days 1, 2 and 3 Doxorubicin 35 mg/m2 IV on Day 1 Cyclophosphamide 1250 mg/m2 IV over 60 minutes on Day 1 Vincristine 1.4 mg/m2 (maximum 2 mg) IV on Day 8 Procarbazine 100 mg/m2 (rounded to nearest 50 mg) orally on Days 1-7 Prednisone 40 mg/m2 (rounded to nearest 5 mg) orally on Days 1-14
Arm/Group | Only Initial Treatment (ABVD x2 Cycles) | Treatment (ABVD:4 Cycles) | Escalated BEACOPP and Involved Field Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/135 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/15 | 12/135 | 2/14
Other Adverse Events (participants affected / at risk) | 8/15 | 131/135 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Only Initial Treatment (ABVD x2 Cycles) (N=15) | Treatment (ABVD:4 Cycles) (N=135) | Escalated BEACOPP and Involved Field Radiation Therapy (N=14)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 5 (5) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 8 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 5 (5) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 3 (3) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
CO diffusing capacity decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 8 (8) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 1 (2) | 7 (7) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Only Initial Treatment (ABVD x2 Cycles) (N=15) | Treatment (ABVD:4 Cycles) (N=135) | Escalated BEACOPP and Involved Field Radiation Therapy (N=14)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 66 (169) | 7 (16)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 7 (7) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (4) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 4 (5) | 1 (3)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 11 (18) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 69 (134) | 5 (9)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 19 (28) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 17 (28) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 29 (45) | 7 (11)
Nausea (Gastrointestinal disorders) | 4 (9) | 111 (288) | 10 (31)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 6 (8) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 2 (5) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 4 (6) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3) | 46 (72) | 5 (9)
Chills (General disorders) | 0 (0) | 5 (8) | 3 (4)
Edema face (General disorders) | 1 (1) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 9 (16) | 1 (1)
Fatigue (General disorders) | 5 (10) | 92 (235) | 9 (23)
Fever (General disorders) | 0 (0) | 17 (23) | 3 (4)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 2 (2) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 3 (4) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 6 (9) | 0 (0)
Localized edema (General disorders) | 0 (0) | 2 (2) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 9 (14) | 3 (4)
Pain (General disorders) | 1 (1) | 10 (13) | 2 (2)
Allergic reaction (Immune system disorders) | 0 (0) | 3 (3) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0/0 (0) | 1 (1) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Phlebitis infective (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (3) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 4 (5) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 9 (9) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 0 (0) | 1 (4) | 0 (0)
Activated partial throm time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 36 (81) | 6 (8)
Alkaline phosphatase increased (Investigations) | 1 (1) | 7 (10) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 29 (57) | 4 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (4) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 4 (4) | 0 (0)
CO diffusing capacity decreased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 3 (3) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Hemoglobin increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 2 (4) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (4) | 28 (53) | 5 (10)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (11) | 113 (337) | 9 (24)
Platelet count decreased (Investigations) | 2 (2) | 9 (10) | 8 (10)
Weight gain (Investigations) | 0 (0) | 8 (14) | 0 (0)
Weight loss (Investigations) | 0 (0) | 3 (3) | 0 (0)
White blood cell decreased (Investigations) | 6 (11) | 112 (334) | 12 (33)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 19 (35) | 3 (7)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 40 (95) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 17 (27) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 12 (19) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 4 (7) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 12 (24) | 4 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 14 (18) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 15 (24) | 4 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 11 (13) | 2 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (10) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 21 (44) | 2 (6)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 19 (39) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 15 (19) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 9 (23) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 26 (37) | 6 (12)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
Olfactory nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 4 (6) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4) | 57 (121) | 5 (10)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (4) | 23 (43) | 4 (9)
Depression (Psychiatric disorders) | 0 (0) | 7 (17) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 18 (39) | 6 (11)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (9) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 44 (66) | 4 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 38 (66) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (13) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (11) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 47 (99) | 3 (5)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 15 (23) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 17 (30) | 1 (2)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 4 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (12) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 2 (5) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 7 (9) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 4 (5) | 1 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 4 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less